CLINICAL TRIAL: NCT02356393
Title: The Effect of Magnesium Serum Levels on Clinical Outcomes in Patients With Acute Myocardial Infarction by Considering Desalination Drinking Water Levels Patients Fed From.
Brief Title: Serum Magnesium Levels in Desalination Tap Water and Outcomes in Acute Myocardial Infarction Patients
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Environment and Health Fund (EHF) (Other)
Responsible Party: Sponsor
Other Study IDs: SHEBA-14-1545-MS-CTIL
Record Dates: First submitted 2014-12-04; First posted 2015-02-05 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Myocardial Infarction; Death; Congestive Heart Failure; Acute-MI; Cardiovascular Disease
Keywords: Desalinated Sea Water; Magnesium; Drinking Water
MeSH Terms: conditions — Myocardial Infarction; Death; Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Association between serum magnesium and clinical outcome in patients with acute MI (AMI) with 1 year follow-up in 300 patients in regions supplied by desalinated drinking water (DSW) (Sheba MC) and 150 patients in regions with non-desalinated drinking water (DW) (Nahariya MC).

DETAILED DESCRIPTION:
Extensive seawater desalination in Israel may decrease magnesium in drinking water (DW), causing hypomagnesemia and adverse health effects. We study the association between consumption of desalinated drinking water (DSW) and serum magnesium in acute MI (AMI) patients, Subjects 35-75 years of age with the first AMI will be prospectively recruited during 1 year from 2 regions; the Departments of Cardiology at the Sheba Medical center (300 patients, predominantly served by DSW) and the Nahariya Medical Center (150 patients, served by non-DSW). Questionnaire will be developed to collect data on demographic variables (at home and work), water and beverages consumption habits (tap water, mineral water), dietary sources of Mg and Mg supplementations. Mg levels will be measured in DW from the patients' homes and in their serum on admission.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with first AMI
2. Age 35-75

Exclusion Criteria:

1. Patients > age 75

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Subjects 35-75 years of age with the first AMI will be prospectively recruited during 1 year from 2 regions; the Departments of Cardiology at the Sheba Medical center (300 patients, predominantly served by DSW) and the Nahariya Medical Center (150 patients, served by non-DSW).
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-05; Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Number of Major Adverse Cardiovascular Events (MACE) | 1 year
  MACE including: acute infarct returns, revascularization, death within 30 days or one year, hospitalization for heart failure, hospitalization for angina pectoris and transient ischemic events.

SECONDARY OUTCOMES:
Age | 1 year
  Age at the first Acute Myocardial Infraction

CONTACTS AND LOCATIONS:
Overall Officials: Meital Shlezinger, PhDcandidate, Study Chair — Haim Sheba medical Center
Locations (1):
- Leviev Heart Center, Chaim Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No